CLINICAL TRIAL: NCT04664309
Title: Understanding Immunity to the COVID-19 Vaccines
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Kari Christine Nadeau, MD, PhD, Professor of Medicine, Stanford University
Other Study IDs: IRB-60171
Record Dates: First submitted 2020-12-09; First posted 2020-12-11 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: COVID-19; Immunity; Vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, saliva, nasal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Adults who are receiving a COVID-19 vaccine
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The purpose of this study is to test over time immunity to the COVID-19 vaccines. Adults who are receiving COVID-19 vaccines will be invited to participate.

ELIGIBILITY:
Inclusion Criteria:

* Adults who are receiving a COVID-19 vaccine

Exclusion Criteria:

* Patients with special risks attendant to venipuncture

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults (18 years and older) receiving a COVID-19 vaccine
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-01-06 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with immunity to COVID-19 vaccines over time | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kari Nadeau, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Hospital, and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No